CLINICAL TRIAL: NCT02200588
Title: A Longitudinal Long-term Study (10 Years) of the Sample of First Episode of Non-affective Psychosis Individuals Included in the First Episode Psychosis Clinical Program (PAFIP)
Brief Title: Longitudinal Long-term Study (10 Years) of the Sample of First Episode of Non-affective Psychosis: PAFIP
Acronym: 10PAFIP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Associate Professor of Psychiatry, Fundación Marques de Valdecilla
Other Study IDs: 10PAFIP
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Schizophrenia
Keywords: psychosis; schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Biospecimen Retention: Samples With DNA — Whole blood, plasma and serum.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients followed in the First Episode Psychosis Clinical Program (PAFIP) with psychotic disorder
- Controls: Healthy subjects without psychotic disorder

SUMMARY:
Schizophrenia is a chronic brain disease that is still understood as a condition that limits the development of a normal life for the patient who suffers it and their families. The idea that only one third of patients have a good outcome is still in force, despite the lack of clinical and epidemiological longitudinal studies that have addressed this issue rigorously. Most studies that have established the poor prognosis of the disease have followed a cross-sectional design and are based on samples of patients undergoing treatment in healthcare devices and therefore represents an important bias. Based on clinical, cognitive, functional outcome and biomarkers studies (brain imaging) to medium term (3 years) we can establish that the particular idea of poor prognosis should be reconsidered. The development of longitudinal studies of first-episode patients in representative samples of a population and long-term it is of high value to shed light on the clinical course of the disease. The belief that there are factors determining the disease progression beyond the initial three years brings us to publish this study.

Given this background, our project's main objective is to know the evolution at 10 years of patients followed in the First Episode Psychosis Clinical Program (PAFIP). Our hypothesis is that a higher percentage of expected patients have a favorable outcome of the disease. Factors such as enhancing treatment completion, abstinence from drug use, return to work, the reduction of expressed emotion in families during the early years of the disease (at least 3 years of intensive intervention PAFIP) will have a positive impact on the evolution of patients on long-term (10 years). Our hypothesis defends the existence of certain factors as independent risk factors for poor clinical and functional outcome of patients who should be known for establishing intervention strategies that attempt to mitigate their impact on the quality of life of patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in the First Episode Psychosis Clinical Program (PAFIP) from February 2001 to December 2007.
* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria of brief psychotic disorder, schizophreniform disorder, schizophrenia or schizoaffective disorder.

Exclusion Criteria:

* Meeting DSM-IV criteria for drug dependence.
* Meeting DSM-IV criteria for mental retardation.
* Having a history of neurological disease or head injury.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals included in the First Episode Psychosis Clinical Program (PAFIP) at the University Hospital Marqués de Valdecilla (Santander - Cantabria).
Sampling Method: Non-Probability Sample
Enrollment: 277 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | At 10 years
  Measured by Disability Assessment Scale (DAS), Global Assessment Functioning (GAF), Quality of Life Scale (QLS), Subjective Well-being under Neuroleptic Scale (SWN-K) and Strauss-Carpenter Scale.

SECONDARY OUTCOMES:
Relapse rate | At 10 years
Change in psychopathology | At 10 years
  Measured by the Scale for the Assessment of Negative and Positive Symptoms (SANS and SAPS), Brief Negative Symptom Scale (BNSS), Brief Psychiatric Rating Scale (BPRS), Clinical Global Impression (CGI-S), Calgary Depression Scale (CDS) and Young Mania Rating Scale (YMRS).
Hospital admission | At 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, Santander, Spain. CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Madrid, Spain
Locations (1):
- University Hospital Marques de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mayoral-van Son J, Juncal-Ruiz M, Ortiz-Garcia de la Foz V, Vazquez-Bourgon J, Setien-Suero E, Tordesillas-Gutierrez D, Gomez-Revuelta M, Ayesa-Arriola R, Crespo-Facorro B; PAFIP Research Group. Long-term clinical and functional outcome after antipsychotic discontinuation in early phases of non-affective psychosis: Results from the PAFIP-10 cohort. Schizophr Res. 2021 Jun;232:28-30. doi: 10.1016/j.schres.2021.04.011. Epub 2021 May 16. No abstract available. PMID 34004383